CLINICAL TRIAL: NCT04657380
Title: A Mobile Application to Improve Case-management and Patient's Functioning in First Episode Psychosis : an Open-label, Multicentre, Superiority, Randomised Controlled Trial Study
Brief Title: A Mobile Application to Improve Case-management and Patient's Functioning in First Episode Psychosis
Acronym: PLAN-e-PSY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PHRCI19FH
Record Dates: First submitted 2020-12-01; First posted 2020-12-08 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Psychosis; Episode
Keywords: FEP; case management; smartphone application; User-centered design; Mixed method; RCT
MeSH Terms: conditions — Psychotic Disorders | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Our hypothesis is that the use of a mobile case-management application for planning and monitoring individualised care objectives, co-designed with patients, their carers, and health professionals, improves the functioning of patients managed for a first psychotic episode, compared to usual case management practices
Who Masked: Outcomes Assessor
Masking Description: Randomisation 1/1 comparing an early intervention program "standard "and an" extended "program within a specialized team will be carried out by IWRS (ENNOV Clinical solution) using the swapped block method. A stratification will be carried out on the case-manager. There is no blinding for the patient or the case-manager. Nevertheless, the evaluation of the comparative outcomes between the 2 groups will be carried out by a psychiatrist who is not involved in the patient's follow-up and who will be blinded to the patient's group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual case management practices (Active Comparator): The first-episode psychosis services participating in the study offer case-management, which will correspond to the treatment as usual in the control group. All the centers are part of the National Transition Network (https://idpsy.org/reseau-transition/centres/). Involvement in this network ensures homogeneity of the usual practices which correspond to the internationally standards. Care delivery is based on intensive treatment during the critical period of psychosis, relying on a wide network of caring and non-caregiving professionals, working together with a view to the successful recovery of the patient. The patient and his or her family are at the center of care and receive proposals for psychoeducation and support throughout the different phases of the illness. This is concomitant with a regular evaluation of patients in order to update the care offer according to their clinical needs.
  Interventions: Behavioral: Control Group
- Mobile case-management application (Experimental): The intervention tested will be a mobile application used during consultations involving the patient and the case manager to define care objectives. The mobile application to be evaluated will result from the process of a co-design phase based on the iterative "user-centered design" approach, involving representatives of carers, patients and caregivers. These stakeholders will define the content and form of the smartphone application during co-building workshops.
  The main purpose of the final application will be to assist in the definition of patients' goals using an approach rooted in recovery theory, with the monitoring of goal achievement in three phases : 1) defining priorities for the patients, through a recovery oriented discussion with the patient and the case manager 2) Setting the concrete objectives and list concrete actions tho achieve them 3) evaluating the achievements.
  Interventions: Behavioral: PLAN-e-PSY mobile application

INTERVENTIONS:
Behavioral: PLAN-e-PSY mobile application — The full version of the application to be evaluated will result from the process of co-design phase of the intervention based on the iterative "user-centered design" approach, involving representatives of carers, patients and caregivers, to define the content and form of the smartphone application during co-building workshops
  Arms: Mobile case-management application
Behavioral: Control Group — The first-episode psychosis services participating in the study offer case-management, which will correspond to the treatment as usual in the control group. All the centers are part of the National Transition Network (https://idpsy.org/reseau-transition/centres/). Involvement in this network ensures homogeneity of the usual practices which correspond to the internationally standards. Care delivery is based on intensive treatment during the critical period of psychosis, relying on a wide network
  Arms: Usual case management practices

SUMMARY:
First Episode Psychosis (FEP) includes perceptual distortions, delusions and cognitive impairment with severe consequences, such as suicidal behaviour. It affects 3% of the population, mainly adolescents and young adults, the majority of with progress to a psychotic disorder.

The early stages of psychotic disorders, from the first full blown symptoms to the next two to five years, represent an opportunity to targeted care and prevention. Indeed, it is a critical period with a worsened clinical prognostic when intervention is delayed, increasing the duration of untreated psychosis (DUP). Also, it is a key period to reduce mortality, as it is characterized by elevated risks of suicide and low physical health outcomes. Besides the symptomatic components, this period is also critical for self-building on educational, professional and emotional levels.

Early intervention programmes involve multi-disciplinary teams, including a care coordination function, embodied by a "case manager". His missions include assessing the patient's needs, developing a care plan to meet the latter, organising access to the different components of the care plan, monitoring and evaluating care, and providing clinical follow-up.

Engagement in the care process is fragile in psychotic disorders, particularly in the context of first episode psychosis with a high risk of care disengagement, often associated with a relapse. It is therefore essential that case-managers involved in FEP services have access to tools designed according to the patient needs and not solely to symptoms, in a "recovery oriented" approach, to foster the feeling of commitment of patients in their care process.

The use of mobile applications for smartphones represents an interesting perspective to improve the engagement of patients with FEP in care. However, the use of an application focused on recovery is feasible and acceptable in patients with first episode psychosis enrolled in a specialised outpatient department (FEP-type service) and allows improvement on clinical criteria, such as psychotic symptoms or mood.

User-centred design methods including identification of users and an inventory of their needs, prototyping with rapid iterations, is a simplification of the procedure and exploitation of existing constraints to increase the rate of use. Moreover, it has recently been shown that such a methodology is feasible in populations with a first episode of psychosis.

Our hypothesis is that the use of a mobile case-management application for planning and monitoring individualised care objectives, co-designed with patients, their careers, and health professionals, improves the functioning of patients managed for a first psychotic episode, compared to usual case management practices.

The originality of our project is built up on two pillars :

* the use of a a mobile monitoring application, which will be used jointly by patients and case-managers,
* the methodological innovation also lies in the collaborative and patient-centred design of the application The originality of our project concerns on the one hand the intervention, an application mobile follow-up, which will be used jointly by patients and case managers. The innovative character also lies at the methodological level in the collaborative and patient-centered design of the application ('user-centered design' approach).

DETAILED DESCRIPTION:
Psychosis and early intervention First Episode Psychosis (FEP) includes perceptual distortions, delusions and cognitive impairment with severe consequences, such as suicidal behaviour. It affects 3% of the population, mainly adolescents and young adults, the majority of wish progress to a psychotic disorder.

From the first full blown symptoms to the next two to five years, the early stages of psychotic disorders represent an opportunity to targeted care and prevention. Indeed, it is a critical period with a worsened clinical prognostic when intervention is delayed, increasing the duration of untreated psychosis (DUP). Also, it Is a key period to reduce mortality, as it is characterized by elevated risks of suicide and low physical health outcomes. Besides the symptomatic components, this period is also critical for self-building on educational, professional and emotional levels.

A pejorative evolution can be avoided by the establishment of "early intervention in psychosis" (EIP), constituted by a set of integrated supports that allow to reduce the symptoms of the disease, promote recovery, foster better social and professional functioning. Moreover, it has recently been shown that EIP reduces general mortality including by suicide in the population monitored. In addition, medico-economic benefits of early intervention have been demonstrated in terms of direct and indirect costs. Thus, this intervention model is currently considered as the reference care in early intervention.

Case management: a strategy to promote recovery in early psychosis Early intervention programmes involve multi-disciplinary teams, including a care coordination function embodied by a "case manager". His missions include assessing the patient's needs, developing a care plan to meet the latter, organising access to the different components of the care plan, monitoring and evaluating care, and providing clinical follow-up. Those missions are broken down into several actions, the content is adapted to the duration of care according to the severity of the disorder and the level of remission.

Case management require essential qualities/ skills such as: accessibility, flexibility, optimism and competence. This model of intervention is effective for patients with FEP and is now considered as a "standard" of care for this population Psychosis and engagement in healthcare: a critical situation In psychotic disorders, the engagement in the care process is fragile, particularly in the context of first episode psychosis with a high risk of care disengagement, often associated with a relapse. Between 20 and 40% of patients with FEP disengage with care despite significant therapeutic needs. The relapse rate one year after stopping treatment ranges from 28% ( to 67% after a first episode of psychosis. Due to the complexity of factors involved in the engagement, it remains endlessly threatened despite better engagement rates in dedicated FEP services compared to "traditional/usual" care, of which the most important is the perception that the service is not adapted to their needs. It is therefore essential that case-managers involved in FEP services have access to tools designed according to the patient needs and not solely to symptoms, in a recovery-oriented approach, to foster the feeling of commitment of patients in their care process.

Mobile applications in mental health: a promising way to promote engagement in FEP services The use of mobile applications for smartphones represents an interesting perspective to improve the engagement of patients with FEP in care. Mobile mental health applications offer many possibilities: an appointment management, an information on the illness, a monitoring of symptoms, a deployment of psychotherapeutic techniques, etc… Mobile applications appear now as promising tools not only for better engagement in care, but also for better self-management capabilities and better coordination of resources. Recent data show an increase in the rate of smartphone equipment in the population of patients with psychosis (over 80%). Qualitative studies in this population show that this type of tools is in great demand, in particular to promote the bound between the patient and services and strengthen the self-management capacities.

Many of the recently implemented applications are aimed for in-patients with short evaluation periods, which does not allow longer term usage data. However, the use of an application focused on recovery is feasible and acceptable in patients with first episode psychosis enrolled in a specialised outpatient department FEP-type service) and allows improvement on clinical criteria, such as psychotic symptoms or mood.

Despite the fact that some applications specifically designed for FEP patients exist and have shown promising results, none have been developed in French and evaluated in French healthcare system. Moreover, anchoring the design of the application in recovery theory would make it possible to better align the actions resulting from the use of the application with the patient's needs.

User-centred design: a method suitable to build "recovery-oriented" tools User-centred design methods, initially developed for human-computer interactions are generally broken down into several phases, including identification of users and an inventory of their needs, prototyping with rapid iterations (i.e. a trial-and-error type strategy allowing rapid feedback from users), simplification of the procedure and exploitation of existing constraints to increase the rate of use. These approaches are particularly developed in the field of mobile application design because they make it possible to create a product that is closer to the concerns of the target person and is so particularly suitable for a "recovery-oriented" approach. Moreover, it has recently been shown that such a methodology is feasible in populations with a first episode of psychosis.

Research hypothesis Our hypothesis is that the use of a mobile case-management application for planning and monitoring individualised care objectives, co-designed with patients, their careers, and health professionals, improves the functioning of patients managed for a first psychotic episode, compared to usual case management practices

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 18 and 30 years old enrolled in a specialised FEP service for a first psychotic episode, defined as follows:

Presence of daily psychotic symptoms for more than a week that have been characterised at the clinical examination by a psychiatrist, Initiation of antipsychotic treatment for less than 6 months, A diagnosis of schizophrenia, schizoaffective disorder, schizophreniform disorder or brief psychotic disorder established according to DSM-5 criteria.

* Mastery of the French language (read and spoken)
* Owning a smartphone
* Adult patients who have given written consent

Exclusion Criteria:

* Patients in psychiatric intensive care units because of severe agitation/disorganisation.
* Patients under guardianship

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 168 (Estimated)
Dates: Start 2022-12-04 (Estimated); Primary Completion 2024-01-04 (Estimated); Study Completion 2025-01-04 (Estimated)

PRIMARY OUTCOMES:
Personal and Social Performance (PSP) scale | Between inclusion and 12 months
  Variation in the patient's functioning score measured by the "Personal and Social Performance (PSP)" scale, informed by a psychiatrist, trained in the use of the scale, not directly involved in the patient's follow-up and blinded to the patient's randomisation group.
  This hetero-evaluative scale, available in French, assesses functioning in a single score that takes into account four domains: productive social activities (work/study), social network, personal care, and disruptive or aggressive behaviour. The integrative score ranges from 0 to 100, with higher scores reflecting better functioning.
  Functioning corresponds to an individual's capacity to assume his or her social role, in the domestic, professional or school, emotional, family and friendship spheres. This is the final objective of case-managed FEPs.

SECONDARY OUTCOMES:
Evolution of the Personal and Social Performance Scale PSP | Between inclusion and 6 months and between inclusion and 12 months
  Evolution of the functioning score measured by the PSP in the patient. The outcome will be the evolution of the PSP score compared in both groups. Total score range: 1 to 100, higher score indicates better functioning.
Therapeutic alliance | Between inclusion and 6 months and between inclusion and 12 months
  Therapeutic alliance as measured by the working alliance inventory (WAI) ): total score range: 36 to 252, higher score indicates better working alliance, patient scale and caregiver scale (case-manager). The outcome will be the evolution of the WAI score compared in both groups.
Adherence to drug treatment | Between inclusion and 6 months and between inclusion and 12 months
  Adherence to drug treatment as measured by the Medical Adherence Rating Scale (MARS) score total score range: 0 to 10, higher score indicates better medical adherence. The assessment criterion will be the evolution of the MARS score compared in both groups.
Psychotic symptomatology | Between inclusion and 6 months and between inclusion and 12 months
  Psychotic symptomatology assessed by the Positive and Negative Symptoms Scale (PANSS) : total score range: 30 to 210, higher score indicates worse symptomatology. This questionnaire hetero assessment gives 3 scores, positive symptoms, negative symptoms and general psychopathology. The outcome will be the evolution of the PANSS score compared in both groups
Recovery | Between inclusion and 6 months and between inclusion and 12 months
  Recovery assessed by the Stages of Recovery Instrument (STORI) the scale is composed of 50 items, grouped in 10 categories. Each categories represents one of the four process components of recovery: hope; identity; meaning; responsibility. The assessment criterion will be the evolution of the STORI score compared in both groups
Life self-report scale | Between inclusion and 6 months and between inclusion and 12 months
  Quality of life assessed by the Schizophrenia Quality of Life self-report scale - 18 items (S-QoL-18) : the scale is composed of 18 items regrouped in 8 dimensions ranging from 0 to 100. A total score is also calculated (range 0-100). Lower scores indicate lower quality of life. The outcome will be the evolution of the S-QoL-18 score compared in both groups
Level of empowerment | Between inclusion and 6 months and between inclusion and 12 months
  Level of empowerment assessed by the Patient Activation Measure (PAM) self-questionnaire (total score range: 0 to 100, higher score indicates higher activation level). The evaluation criterion will be the evolution of the PAM score compared in both groups.
Patient engagement in care | Between inclusion and 6 months and between inclusion and 12 months
  Patient engagement in care assessed by the Service Engagement Scale (SES) translated into French (: total score range: 0 to 42. Higher scores reflected clients' greater levels of difficulty engaging with services). The evaluation criterion will be the evolution of the SES score compared in both groups.
Patient satisfaction with case-management | Between inclusion and 6 months and between inclusion and 12 months
  Patient satisfaction with case-management assessed by a self-administered questionnaire constructed in the study using a visual analogue scale (VAS). The evaluation criterion will be the evolution of the VAS score compared in the centre and both groups
Hospitalisation for relapse of psychosis | Over12 months
  Evaluation in the patient in both groups of the number of days of hospitalisation for relapse of psychosis, collected at follow-up.
Acceptability and appropriation of the PLAN-e-PSY application | At 12 months
  The acceptability and appropriation of the application (intervention group) by patients (strengths and limitations of the application) and the case-manager (strengths and limitations of the application, perceived change in practices, commitment) assessed during the semi-structured interviews
Fidelity of use of the PLAN-e-PSY application | Over12 months
  Fidelity of use by the case manager and patients of the different parts of the application in relation to the defined procedures. These elements will be collected from the application's internal monitoring data
Case manager effective use of the PLAN-e-PSY application | At 12 months
  Proportion of case manager consultations during which the application was not used. These elements will be collected from the application's internal monitoring data
Patient effective use of the PLAN-e-PSY application | At 12 months
  Proportion of patients who stopped using the application. These elements will be collected from the application's internal monitoring data
Time of effective use of the PLAN-e-PSY application | Over 12 months
  Time of effective use by the case manager and patients of the application. These elements will be collected from the application's internal monitoring data

CONTACTS AND LOCATIONS:
Overall Officials: Frederic HAESEBAERT, PH, Principal Investigator — Centre Hospitalier le Vinatier
Locations (1):
- Ch Le Vinatier, Lyon, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Haesebaert F, El Oussoul S, Pavard A, Fabre D, Cellard C, Magaud L, Subtil F, Damiolini E, Fakra E, Haesebaert J. PLAN-e-PSY, a mobile application to improve case management and patient's functioning in first episode psychosis: protocol for an open-label, multicentre, superiority, randomised controlled trial. BMJ Open. 2021 Sep 14;11(9):e050433. doi: 10.1136/bmjopen-2021-050433. PMID 34521670